CLINICAL TRIAL: NCT00625612
Title: A Phase 3, International, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Efficacy and Safety Study of Denufosol Tetrasodium Inhalation Solution in Patients With Cystic Fibrosis Lung Disease and FEV1 Greater Than or Equal to 75% Predicted But Less Than or Equal to 110% Predicted
Brief Title: Study of Denufosol Tetrasodium Inhalation Solution in Patients With Cystic Fibrosis (CF) Lung Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P08640; 08-110
Record Dates: First submitted 2008-02-12; First posted 2008-02-28 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — denufosol tetrasodium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo
- 1 (Experimental): Denufosol Tetrasodium (INS37217) Inhalation Solution
  Interventions: Drug: Denufosol Tetrasodium (INS37217) Inhalation Solution

INTERVENTIONS:
Drug: Denufosol Tetrasodium (INS37217) Inhalation Solution — Drug: Denufosol Tetrasodium (INS37217) Inhalation Solution, Denufosol 60 mg is administered as an inhalation solution, three times daily for twelve months.
  Arms: 1
Drug: Placebo — Placebo - 0.9% w/v sodium chloride solution, three times daily for twelve months.
  Arms: 2

SUMMARY:
The purpose of this trial is to evaluate the safety and effectiveness of one dose strength of Denufosol compared to placebo in patients with CF and a predicted FEV1 of greater than or equal to 75% but less than or equal to 110% predicted.

ELIGIBILITY:
Inclusion Criteria:

* Have confirmed diagnosis of cystic fibrosis
* Have FEV1 of greater than or equal to 75% but less than or equal to 110%predicted normal for age, gender and height
* Be able to reproducibly perform spirometry
* Be clinically stable for at least 4 weeks before screening

Exclusion Criteria:

* Have abnormal renal or liver function
* Have lung transplant
* Unable to discontinue use of hypertonic saline
* Participated in Inspire trial 08-108

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 466 (Actual)
Dates: Start 2008-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Change in lung function | 48 weeks

SECONDARY OUTCOMES:
Pulmonary Exacerbation, Antibiotic Use, Incidence of Hospitalization/ER visits, Health resource utilization, Quality of Life | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Felix Ratjen, MD, PhD, Principal Investigator — Toronto, Canada
Locations (105):
- United States (82):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Pediatric Breathing Disorders, Anchorage, Alaska
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - University of Arizona/Arizona Health Sciences, Tucson, Arizona
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - USC Cystic Fibrosis Center, Los Angeles, California
  - Bay Area Pediatric Pulmonary, Oakland, California
  - Kaiser Permanente Medical Center, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Sanford University, Palo Alto, California
  - Capital Allergy & Respiratory Disease Center, Sacramento, California
  - UCSD Medical Center - Hillcrest & Thornton Hospitals, San Diego, California
  - UCSD Medical Center - Hillcrest and Thornton Hospitals, San Diego, California
  - Pediatric Diagnostic Center, Ventura, California
  - Yale School of Medicine, New Haven, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Shands at University of Florida, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Nemours Children's Clinic, Pensacola, Florida
  - Pediatric Pulmonary Associates, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - St. Mary's Medical Center, West Palm Beach, Florida
  - Emory University, Atlanta, Georgia
  - Children's Healthcare of Atlanta at Scottish Rite, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - Cystic Fibrosis Institute, Glenview, Illinois
  - James Whitcomb RIley Hospital for Children, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Via Christa Research, Wichita, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Tulane University Medical Center, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - Children's Health Care, Minneapolis, Minnesota
  - University of Minnesota - Farview, Minneapolis, Minnesota
  - Childrens Mercy Hospital, Kansas City, Missouri
  - Saint Louis University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Children's Lung Specialists, Las Vegas, Nevada
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - The Respiratory Center for Children, Morristown, New Jersey
  - Albany Medical College, Albany, New York
  - Cystic Fibrosis Center of Schneider Children's Hospital, Great Neck, New York
  - New York Medical College, Hawthorne, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - St. Vincent's Catholic Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Duke University Medical Center, Durham, North Carolina
  - St. Alexius Medical Center, Bismarck, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospital of Cleveland, Cleveland, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - The Children's Medical Center of Dayton, Dayton, Ohio
  - Toledo Children's Hospital, Toledo, Ohio
  - Santiago Reyes, MD, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - PennState Milton S Hershey Med, Hershey, Pennsylvania
  - The Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Childrens Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Sanford Childrens' Specialty Clinic, Sioux Falls, South Dakota
  - East Tennesse Children's Hospital - Pediatric Pulmonary and Respiratory Care, Knoxville, Tennessee
  - Austin Children's Chest Associates, Austin, Texas
  - Dallas Cystic Fibrosis Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Naval Medical Center Portsmouth, Portsmouth, Virginia
  - Pediatric Pulmonary Clinic, Richmond, Virginia
  - West Virginia University, Morgantown, West Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - University of Wisconsin School of Medicine and Pulbic Health, Madison, Wisconsin
- Australia (11):
  - John Hunter Hospital - Adults, New Lambton, New South Wales
  - Westmead Adults, Westmead, New South Wales
  - Prince Charles Hospital, Chermside, Queensland
  - Royal Brisbane Children's Hospital, Herston, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Respiratory Medicine, Parkville, Victoria
  - Sire Charles Gairdner Hospital, Nedlands, Western Australia
  - Princess Margaret Hospital for Children, Perth, Western Australia
  - The Children's Hospital of Westmead, Westmead
- Canada (11):
  - University of Calgary, Alberta Children's Hospital, Calgary, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Eastern Health, St. John's, Newfoundland and Labrador
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - McMaster University, Hamilton, Ontario
  - A. Lyttle Research COmpany, London, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - University of Toronto, Toronto, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Centre Mere-Enfant du CHUL, Montreal, Quebec
- Green Lane Clinical Centre (NZ), Auckland, New Zealand

REFERENCES:
- [Derived] Ratjen F, Durham T, Navratil T, Schaberg A, Accurso FJ, Wainwright C, Barnes M, Moss RB; TIGER-2 Study Investigator Group. Long term effects of denufosol tetrasodium in patients with cystic fibrosis. J Cyst Fibros. 2012 Dec;11(6):539-49. doi: 10.1016/j.jcf.2012.05.003. Epub 2012 Jun 8. PMID 22682898